CLINICAL TRIAL: NCT05007314
Title: Biocriminology and the Adjudication of Criminal Responsibility: Is There a Consensus Among Scientists' Verdicts?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Mia Athina Thomaidou, Principal Investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2021-07-16-D.S.V.-V2-3332
Record Dates: First submitted 2021-08-02; First posted 2021-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Criminalism
Keywords: Punishment; Responsibility; Attitudes
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human Science (Experimental): Arm 1 will include university graduates that hold at least a science undergraduate degree (or equivalent) in human science, including psychology, neuroscience, human biology, or medicine.
  Interventions: Behavioral: Biocriminological Evidence
- Natural or non-science (Active Comparator): Arm 2 will include university graduates from non-human or non-scientific fields such as engineering, history, language studies, or law.
  Interventions: Behavioral: Biocriminological Evidence

INTERVENTIONS:
Behavioral: Biocriminological Evidence — Participants in each of the two main groups see a case with and a case without a neurobiological explanation for criminal offending.

SUMMARY:
Because of the evolving nature of psychology research, non-scientists are more likely to struggle or misinterpret evidence regarding a person's psychological state. Misconceptions may thus be highly prevalent within the justice system, leading to negative consequences for people with psychological or neurobiological disorders. At the same time, no research has been conducted to compare the punishment perspectives of non-scientists, that typically make sentencing decisions, to scientists who possess a more advanced understanding of human biology and behavior.

DETAILED DESCRIPTION:
In this study, closely inspired by the paradigms of Berryessa, Coppola, and Salvato, perspectives on punishment based on psychobiological explanations of behaviour are assessed, aiming to understand how scientists with knowledge of human psychobiology versus lay people (of similar educational level) interpret offending behaviour. Human-science is contrasted to natural-science/arts graduates because the former have been exposed to and may possess scientific knowledge that shapes their understanding of behaviour, their views, and potential (essentialist) biases. In contrast, non-scientists have been found to possess scientific misconceptions that can impact their sentencing decisions. This leads to the question whether scientists may draw different judgements based on their professional knowledge and experience with psychological phenomena. If indeed scientists with greater insight on human behaviour are found to hold less punitive views on punishment and rehabilitation, that has important implications for criminal justice systems that rely on lay peoples' understanding of science.

One hundred sixty participants who completed all study procedures (2 main groups of 80 participants) will be surveyed. A sample size calculation was performed using G*Power version 3.1.9.4, based on Berryessa and colleagues who conducted a similar survey study in 2021 with comparable outcome measures and analyses. The required effect size is based upon approximately 3-4 outcome measures. The primary research question is between-groups, while secondary ones include within groups measures. Based on the power analysis, a sample of 160 participants will be targeted, which is enough for sufficient power for f = 0.25, power = 0.80, df = 4, for 2 different groups.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65
* Holding a university diploma or equivalent

Exclusion Criteria:

* Participants who did not complete the survey (appropriately) will be excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Lived gender
Enrollment: 160 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Sentencing severity on 5-point questionnaire | Immediately after case presentation, an average of 1 minute.
  This is the primary outcome measure of attitudes towards sentencing, measured via a questionnaire on a visual analogue scale from 1 (only treatment) to 5 (more than 5 years in prison)

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Raw anonymised data, processing and analysis steps, and all code, will be provided via an online repository or as required by a scientific journal.
Supporting Information: Study Protocol, Analytic Code
Time Frame: After the publication of the study
Access Criteria: For quality assurance and potential use in relevant research when deemed applicable